CLINICAL TRIAL: NCT01792362
Title: Comparing the Basal Anti-mullerian Hormone Levels Between Responders and Non-responders to Weight Loss Diet in Obese Infertile Women With PCOS Population
Brief Title: Evaluation of Anti-mullerian Hormone(AMH) Levels as a Predictive Factor of Response to Weight Loss Treatment in Obese Infertile Women With Poly Cystic Ovary(PCOS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Emb-015
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2012-11

CONDITIONS: Infertility
Keywords: Anti-mullerian hormone (AMH) level, poly cystic ovarian syndrome obese infertility weight loss diet
MeSH Terms: conditions — Infertility | interventions — Diet, Reducing

ARMS (1):
- AMH (Experimental): obese PCOS patients who underwent weight loss diet
  Interventions: Other: Weight loss diet

INTERVENTIONS:
Other: Weight loss diet — Control the patients diet to make them loosing weight

SUMMARY:
This study is a prospective before & after clinical trial to compare the basal and 3 months after diet anti-mullerian hormone levels between responders and non-responders to weight loss diet in obese infertile women with PCOS population

DETAILED DESCRIPTION:
The study population comprised of all obese infertile PCOS patients aged 20-40 years which underwent 3 months weight loss diet in royan institute, Tehran Iran.

The study is conducted over 12 wk energy restriction. All subjects have the same dietary protocol. At baseline, week 12 the levels of AMH,Follicular Stimulating Hormone (FSH), Lutienizing Hormone(LH),Prolactin (PRL), androgens, sex hormone-binding globulin (SHBG), glucose, and insulin were measured and Free Androgen Index (FAI) and Insulin Resistance (IR) indices is calculated. The laboratory tests are determined by radioimmunoassay in the Laboratory of Endocrinology of Royan institute. AMH is measured in duplicate using an ultrasensitive ELISA kit (AMH-ELIZA Kit; Beckman Coulter, Marseilles, France) according to manufacturer instructions. All measurements are performed using a single kit and at the same time in the Laboratory of clinical Immunology of Royan institute.

Data collection will be performed by using questionnaire to be filled as per the available records and laboratory results. Data analysis will be done through descriptive and perceptive statistical methods.

ELIGIBILITY:
Inclusion Criteria:

- 1- diagnosis of PCOS, according to the Rotterdam Consensus Workshop Group, by 2 of the following 3 criteria: menstrual irregularity (cycle length<26 d or >31 d or variation between consecutive cycles of >3 d); clinical (hirsutism assessed by a Ferriman-Gallwey score > 8) or biochemical [free androgen index (FAI) > 5.4 or testosterone_1.4 nmol/L] hyperandrogenism; or positive ultrasound presentation of polycystic ovaries by transvaginal scan.

2- Age between 18 -40

Exclusion Criteria:

- 1. Body mass index (BMI; in kg/m2) < 30, 2. Type 2 diabetes mellitus and related endocrinopathic disorders [identified by assessment of thyroid-stimulating hormone (TSH), prolactin, and 17_hydroxyprogesterone].

3. Regular exercise activities during the study. 4. Cases of alcoholism and smoking. 5. The use of endocrine hormonal treatment or insulin-sensitizing agents is not permitted during either phase of the study, and the use of oral contraceptives is not permitted during of the study. Subjects are required to cease taking oral contraceptives 4 wk and hormonal treatment or insulin-sensitizing agents 2 wk before commencement of the short-term study phase.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Blood level of AMH | 3 months
  Evaluation of Blood level of AMH 12 weeks after weight loss.
Basal level of AMH | 1 week
  Evaluation the Basal level of AMH before starting weight loss diet

SECONDARY OUTCOMES:
Sensitivity of basal AMH level | 6 months
  Evaluation the Sensitivity of basal AMH level for predict the response to weight loss diet
specificity of basal AMH level | 6 months
  Evaluation the specificity of basal AMH level for predict the response to weight loss diet

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Ashraf Moini, MD, Study Director — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Center, Royan institute for Reproductive Biomedicine, ACECR, Tehran, Iran
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org